CLINICAL TRIAL: NCT02986126
Title: Resilience Against Depression Disparities (Also Known as Resilience Education to Reduce Depression Disparities)
Acronym: RADD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bowen Chung, MD, MSHS (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other); Tulane University (Other); Healthy African American Families II (Unknown); University of California, San Francisco (Other); Arming Minorities Against Addiction & Disease (Unknown); Louisiana Community Health Outreach Network (Unknown)
Responsible Party: Sponsor-Investigator, Bowen Chung, MD, MSHS, Associate Professor-in-Residence, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PPRND-1507-32173
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Depressive Symptoms
Keywords: Depression; Resilience; Minority health; Community-based participatory research; Lesbian, gay, bisexual, transgender, and intersex (LGBTI) health; Racial / ethnic health disparities; Patient-centered outcomes research; Comparative-effectiveness research
MeSH Terms: conditions — Depression; Homosexuality, Female; Homosexuality; Bisexuality; Ovotesticular Disorders of Sex Development | interventions — Health Resources

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resources for Services (Active Comparator): Resources for Services (RS) is an evidence-based depression QI toolkit developed for primary care, but adapted for health- and community-based programs. Protocols support training licensed providers in clinical assessment, medication management, and CBT; all staff in team management; and non-clinical staff in addressing patient safety, screening, behavioral management skills (behavioral activation, problem solving) to enable education, coordination, and referral. RS is offered as an initial 1-day / 8-hour training with follow-up through 12 webinars, 3 each on team management, medication management, psychotherapy, and case management. Programs will be invited to have a staff lead per training component, with no limit on number of staff at trainings. Training experts include a psychiatrist, psychologist/CBT trainer, case manager, support staff, and patient / community advocate liaison. All enrolled study participants will be nested within programs participating in RS.
  Interventions: Other: Resource for Services (RS)
- Resiliency Class + (Active Comparator): Resiliency Classes (RC) are a manualized, 7-session, CBT, psychoeducation class, lead by community health workers, that teaches skills to enhance mood. The RC manual covers: Session 1 - "What Affects Your Mood and Resilience;" Session 2 - "Pleasant Activities Can Help Improve Your Mood and Make You Resilient;" Session 3 - "What Gets In The Way of Pleasant Activities: Harmful Thoughts and How to Change Them;" Session 4 - "How to Increase Your Resilience Through Support from Others;" Session 5 - "My Personal Resiliency Plan: Goal Setting;" Session 6 - "Celebrate Your Resiliency: Graduation" Each RC will be 90-120 minutes in duration; once a week in community settings with up to 10 participants. RC will be supplemented with automated mobile text reminders about basic concepts and follow-up for care. Half of enrolled participants will be randomized to the Resiliency Class +. As of July 12, 2018, we will be offering bus tokens and $5 for completion of a satisfaction survey.
  Interventions: Behavioral: Resiliency Class; Other: Resource for Services (RS)

INTERVENTIONS:
Behavioral: Resiliency Class — See Arm Description
  Arms: Resiliency Class +
Other: Resource for Services (RS) — See Resource for Services (RS) Description
  Other Names: Active Comparator

SUMMARY:
Depressive symptoms and disorders are among the most common adult health conditions with a lifetime prevalence of 15-20% and are a leading cause of disability /morbidity worldwide. Although evidence-based approaches such as cognitive behavioral therapy (CBT), antidepressant medications, and depression collaborative care and quality improvement (QI) programs integrating depression care into primary health care can improve depression outcomes and disparities, racial / ethnic disparities continue to persist. Concurrently, according to a 2011 Institute of Medicine (IOM) report, little information exists on how to address the high rates of depression among sexual and gender minorities.

Our study randomizes depressed, LGBTQ (lesbian, gay, bisexual, transgendered, queer), racial / ethnic minority adults to an evidence-based agency-level, depression quality improvement (QI) training [Resources for Services (RS)] and technical support alone or to a resiliency class (RC+), a 7-session resiliency, cognitive behavioral therapy class to enhance mood + automated mobile text reminders about basic reminders and care follow-up impact on improving adult patients' depressive symptoms. Depression QI (RS) training will be offered to three clusters of four to five LGBTQ-focused programs: two clusters in LA (Hollywood and South LA) and one cluster in NO. Clusters are comprised of one primary care, one mental health, and two to three community agencies (e.g., faith-based, social services/support, advocacy). All programs will receive depression QI training. Enrolled adult depressed patients (n=320) will be randomized individually to RC+ or RS (depression QI) alone to assess effects on primary outcomes: depressive symptoms [8-item patient health questionnaire (PHQ-8) score and secondary outcomes: mental health quality of life [12-item mental composite score (MCS-12) ≤ 40], Resilience (Brief Resilience Scale), mental wellness, and physical health quality of life [12-item physical composite (PCS-12)score] at 6- and 12-month follow-up.

DETAILED DESCRIPTION:
Depressive symptoms and disorders are among the most common adult health conditions and are a leading cause of disability /morbidity worldwide. Although evidence-based approaches such as cognitive behavioral therapy (CBT), antidepressant medications, and depression collaborative care and quality improvement (QI) programs integrating depression care into primary health care can improve depression outcomes and disparities, racial / ethnic disparities continue to persist. Concurrently, according to a 2011 Institute of Medicine (IOM) report notes little information exists on how to address the high rates of depression among sexual and gender minorities, largely composed of lesbian, gay, and bisexual (LGBTQ) individuals. Limited comparative effectiveness data exists to know what treatments and services options improve health disparities due to patient characteristics such as race / ethnicity, and sexual orientation.

"Resilience Against Depression Disparities (RADD)" randomizes enrolled depressed, LGBTQ, racial / ethnic minority adults (n=320) to an agency-level, evidence-based depression quality improvement (QI) intervention [Resources for Services (RS)] training and technical support and then randomizes individuals to Resources for Services alone or to Resiliency Class+, a 7-session resiliency, depression cognitive behavioral therapy class + automated mobile text reminders about basic reminders and care follow-up impact on improving adult patients' depressive symptoms over 6- and 12-months. RS training will be offered to three clusters of four to five LGBTQ-focused programs: two clusters in LA (Hollywood and South LA) and one cluster in NO. Clusters are comprised of one primary care, one mental health, and two to three community agencies (e.g., faith-based, social services/support, advocacy). All programs will receive RS (depression QI training). All enrolled adult depressed patients will be within programs participating in RS (depression QI) trainings. Half of enrolled participants will be randomized to the Resilience Class +.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. moderately to severely depressed (PHQ-8≥10)
3. Able to be contacted by phone (voice or text message), e-mail, or Facebook.
4. English or Spanish speaker

Exclusion Criteria:

1. Under age 18 years
2. Not moderately to severely depressed (PHQ-8≤10)
3. Does not currently have a phone, an email address, or a Facebook profile

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Depressive symptom count as measured by the Patient Health Questionnaire 8 | Change from baseline at 6- and 12-month follow-up
  The 8-item Patient Health Questionnaire (PHQ-8) is a standard measure of depressive symptoms.

SECONDARY OUTCOMES:
Poor Mental Health-Related Quality of Life | 6- and 12-month follow-up
  12-item mental composite score (MCS-12) ≤ 40
Resilience | 6- and 12-month follow-up
  Brief Resilience Scale
Physical health-related quality of life | 6- and 12-month follow-up
  12-item physical composite score (PCS-12)
Mental Wellness | 6- and 12-month follow-up
  3 items in last 4 weeks: some feeling of being calm or peaceful, having energy or being happy (from 36-item Short Form Health Survey)

CONTACTS AND LOCATIONS:
Overall Officials: Bowen Chung, MD, MSHS, Principal Investigator — University of California, Los Angeles
Locations (22):
- United States (22):
  - R.O.A.D.S. Clinic, Compton, California
  - The ADAM Project - YMSM Program, Long Beach, California
  - The LGBTQ Center - Long Beach, Long Beach, California
  - AMAAD, Los Angeles, California
  - AIDS Health Foundation Healthcare Center - Downtown Los Angeles, Los Angeles, California
  - AIDS Health Foundation Healthcare Center - Hollywood, Los Angeles, California
  - AIDS Health Foundation Public Health Division, Los Angeles, California
  - Metropolitan Community Church, Los Angeles, California
  - OASIS Clinic, Los Angeles, California
  - Southern Transmasculine Alliance, New Orleans, Louisiana
  - New Orleans Musicians Clinic, New Orleans, Louisiana
  - St. Anna's Church, New Orleans, Louisiana
  - Crescent Care - The Community Awareness Network (CAN Office), New Orleans, Louisiana
  - Crescent City Sanctuary, New Orleans, Louisiana
  - Metropolitan Community Church of New Orleans, New Orleans, Louisiana
  - NOAGE, New Orleans, Louisiana
  - Brotherhood, New Orleans, Louisiana
  - Crescent Care - The Movement, New Orleans, Louisiana
  - Crescent Care, New Orleans, Louisiana
  - Odyssey Home, New Orleans, Louisiana
  - Sisters of Perpetual Indulgence - The Big Easy Sisters, New Orleans, Louisiana
  - Women with a Vision, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Undecided
We will work with the Patient-Centered Outcomes Research Institute (PCORI) staff as the findings emerge to determine the potential value of some or all of the dataset being made publicly available, which would require additional funding from PCORI to complete. In general PCORI works with investigators to make a complete, cleaned, de-identified final data set with detailed descriptions contained within the study protocol available to PCORI for use as a publicly available dataset after study completion.

REFERENCES:
- [Result] Moussavi S, Chatterji S, Verdes E, Tandon A, Patel V, Ustun B. Depression, chronic diseases, and decrements in health: results from the World Health Surveys. Lancet. 2007 Sep 8;370(9590):851-8. doi: 10.1016/S0140-6736(07)61415-9. PMID 17826170
- [Result] Miranda J, Chung JY, Green BL, Krupnick J, Siddique J, Revicki DA, Belin T. Treating depression in predominantly low-income young minority women: a randomized controlled trial. JAMA. 2003 Jul 2;290(1):57-65. doi: 10.1001/jama.290.1.57. PMID 12837712
- [Result] Wells KB, Sherbourne C, Schoenbaum M, Duan N, Meredith L, Unutzer J, Miranda J, Carney MF, Rubenstein LV. Impact of disseminating quality improvement programs for depression in managed primary care: a randomized controlled trial. JAMA. 2000 Jan 12;283(2):212-20. doi: 10.1001/jama.283.2.212. PMID 10634337
- [Result] Wells KB, Tang L, Miranda J, Benjamin B, Duan N, Sherbourne CD. The effects of quality improvement for depression in primary care at nine years: results from a randomized, controlled group-level trial. Health Serv Res. 2008 Dec;43(6):1952-74. doi: 10.1111/j.1475-6773.2008.00871.x. Epub 2008 Jun 3. PMID 18522664
- [Result] Gilbody S, Bower P, Fletcher J, Richards D, Sutton AJ. Collaborative care for depression: a cumulative meta-analysis and review of longer-term outcomes. Arch Intern Med. 2006 Nov 27;166(21):2314-21. doi: 10.1001/archinte.166.21.2314. PMID 17130383
- [Result] Miranda J, Duan N, Sherbourne C, Schoenbaum M, Lagomasino I, Jackson-Triche M, Wells KB. Improving care for minorities: can quality improvement interventions improve care and outcomes for depressed minorities? Results of a randomized, controlled trial. Health Serv Res. 2003 Apr;38(2):613-30. doi: 10.1111/1475-6773.00136. PMID 12785564
- [Result] Institute of Medicine (US) Committee on Lesbian, Gay, Bisexual, and Transgender Health Issues and Research Gaps and Opportunities. The Health of Lesbian, Gay, Bisexual, and Transgender People: Building a Foundation for Better Understanding. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK64806/ PMID 22013611
- [Result] Springgate BF, Wennerstrom A, Meyers D, Allen CE 3rd, Vannoy SD, Bentham W, Wells KB. Building community resilience through mental health infrastructure and training in post-Katrina New Orleans. Ethn Dis. 2011 Summer;21(3 Suppl 1):S1-20-9. PMID 22352077
- [Result] Wells KB, Jones L, Chung B, Dixon EL, Tang L, Gilmore J, Sherbourne C, Ngo VK, Ong MK, Stockdale S, Ramos E, Belin TR, Miranda J. Community-partnered cluster-randomized comparative effectiveness trial of community engagement and planning or resources for services to address depression disparities. J Gen Intern Med. 2013 Oct;28(10):1268-78. doi: 10.1007/s11606-013-2484-3. Epub 2013 May 7. PMID 23649787
- [Result] Chung B, Ong M, Ettner SL, Jones F, Gilmore J, McCreary M, Sherbourne C, Ngo V, Koegel P, Tang L, Dixon E, Miranda J, Belin TR, Wells KB. 12-month outcomes of community engagement versus technical assistance to implement depression collaborative care: a partnered, cluster, randomized, comparative effectiveness trial. Ann Intern Med. 2014 Nov 18;161(10 Suppl):S23-34. doi: 10.7326/M13-3011. PMID 25402400
- [Result] Chung B, Ngo VK, Ong MK, Pulido E, Jones F, Gilmore J, Stoker-Mtume N, Johnson M, Tang L, Wells KB, Sherbourne C, Miranda J. Participation in Training for Depression Care Quality Improvement: A Randomized Trial of Community Engagement or Technical Support. Psychiatr Serv. 2015 Aug 1;66(8):831-9. doi: 10.1176/appi.ps.201400099. Epub 2015 May 1. PMID 25930037
- [Result] Katon WJ, Lin EH, Von Korff M, Ciechanowski P, Ludman EJ, Young B, Peterson D, Rutter CM, McGregor M, McCulloch D. Collaborative care for patients with depression and chronic illnesses. N Engl J Med. 2010 Dec 30;363(27):2611-20. doi: 10.1056/NEJMoa1003955. PMID 21190455
- [Result] U.S. Department of Health and Human Services. Advancing LGBT Health & Well-Being: 2014 Report. 2014; http://www.hhs.gov/programs/topic-sites/lgbt/index.html.
- [Derived] Vargas SM, Wennerstrom A, Alfaro N, Belin T, Griffith K, Haywood C, Jones F, Lunn MR, Meyers D, Miranda J, Obedin-Maliver J, Pollock M, Sherbourne CD, Springgate BF, Sugarman OK, Rey E, Williams C, Williams P, Chung B. Resilience Against Depression Disparities (RADD): a protocol for a randomised comparative effectiveness trial for depression among predominantly low-income, racial/ethnic, sexual and gender minorities. BMJ Open. 2019 Oct 22;9(10):e031099. doi: 10.1136/bmjopen-2019-031099. PMID 31641001
- See also: Patient-Centered Outcomes Research Institute Project Summary — http://www.pcori.org/research-results/2016/resiliency-education-reduce-depression-disparities